CLINICAL TRIAL: NCT04261335
Title: The Evaluation of Safety and Tolerability of CL2020 in Neonatal Hypoxic Ischemic Encephalopathy Patients With Therapeutic Hypothermia in the Dose Escalation Clinical Trial
Brief Title: The Clinical Trial of CL2020 Cells for Neonatal Hypoxic Ischemic Encephalopathy
Acronym: SHIELD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nagoya University (Other)
Collaborators: Life Science Institute, Inc. (Unknown)
Responsible Party: Principal Investigator, Yoshiaki Sato, MD, PhD, Associate Professor at Department of Center for Maternal Neonatal Care, Nagoya University Hospital, Nagoya University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMCR-014; jRCT2043190112 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2020-02-01; First posted 2020-02-07 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Hypoxia-Ischemia, Brain
Keywords: Hypoxia-Ischemia, Brain; Infant, Newborn; Mesenchymal Stem Cells
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Intervention Model Description: 3 + 3 dose escalation study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CL2020 cells (Experimental): Intravenous injection of CL2020 cells
  Interventions: Biological: CL2020 cells

INTERVENTIONS:
Biological: CL2020 cells — 1.5 million or 15 million cells, IV on day 5 to 14 of birth

SUMMARY:
The purpose of this study is to evaluate the safety and the tolerability of CL2020 cells in hypoxic ischemic encephalopathy neonates with hypothermia therapy. In addition, we will evaluate the efficacy of CL2020 cells for infant development.

ELIGIBILITY:
Inclusion Criteria:

1. At least 36 weeks gestation, and either one of the following criteria (i.-iii.) i. Apgar score ≤5 at 10 minutes ii. Continued resuscitation for at least 10 minutes iii. pH <7.0 or base deficit ≥16 mmol/L in any blood sample obtained within 60 min of birth
2. Moderate or severe encephalopathy by a Sarnat criteria
3. Undergone therapeutic hypothermia started before six hours of birth, and done for 72 hours continuously
4. Birth weight ≥1,800 g
5. Heart rate ≥100/min, and SpO2 ≥90 %
6. Able to provide voluntary written consent after receiving adequate information about the study (consent will be obtained from an acceptable representative)

Exclusion Criteria:

1. Suspected or confirmed severe congenital abnormalities or chromosomal anomaly
2. Planned to undergo surgery or radiation therapy
3. Scheduled to take systemic corticosteroids treatment for over five days
4. Blood glucose ≥ 200 mg/dL
5. Participation in another clinical study (not exclude patients in observational studies)
6. Suspected or confirmed active and severe infection
7. Positive for HBs antigen, HCV antibody, HIV antibody, HTLV-1 antibody or syphilis serum reaction
8. History of severe hypersensitivity or anaphylactic reaction
9. Severe complications

Ages: 4 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | until 12 weeks after the administration
  Any adverse events are summarized.

SECONDARY OUTCOMES:
Incidence of composite endpoints (death, continuous respiratory support, and continuous use of vasopressors or pulmonary vasodilators) | at 12, 26, 38, 52, and 78 weeks after administration
  Incidence of composite endpoints is summarized.
Mortality | all of the clinical trial period (up to 44 months)
  Mortality is summarized.
Overall survival | all of the clinical trial period (up to 44 months)
  Overall survival is summarized.
Duration of continuous respiratory support | up to 78 weeks
  Duration of continuous respiratory support is summarized.
Duration of continuous use of vasopressors or pulmonary vasodilators | up to 78 weeks
  Duration of continuous use of vasopressors or pulmonary vasodilators is summarized.
The composite score of cognitive scale, language scale, motor scale, social-emotional scale, and adaptive behavior scale in Bayley Scales of Infant and Toddler Development Third edition | 78 weeks after administration
  Each composite scores are summarized. The higher scores mean a better outcome.
The developmental quotient in Kyoto Scale of Psychological Development 2001 | 78 weeks after administration
  The developmental quotient is summarized. The higher scores mean a better outcome.
Presence of 1) head control, 2) roll over, 3) sitting position, 4) crawl, 5) independent gait, and 6) meaningful words | at 26, 38, 52, and 78weeks after administration
  Presence of each event is summarized.
Presence of spasticity | at 12, 26, 38, 52, and 78 weeks after administration
  Presence of spasticity is summarized. Spasticity is the condition as below: increased muscle tone, or increased deep tendon reflex.
Presence of epilepsy | until 78 weeks after administration
  Presence of spasticity is summarized. The definition of epilepsy is the condition based on the International League Against Epilepsy.
MRI score | at 2, and 78 weeks after administration
  MRI score is summarized. The scoring system is based on the report of Barkovich AJ, et al. (AJNR Am J Neuroradiol. 1998 ;19(1):143-9.) . The higher scores mean a worse outcome.
Gross Motor Function Classification System (GMFCS) score | at 78 weeks after administration
  GMFCS score is summarized. The gross motor function can be categorized into 5 different level. The higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiaki Sato, MD, PhD, Principal Investigator — Department of Center for Maternal Neonatal Care, Nagoya University Hospital
Locations (1):
- Nagoya University Hospital, Nagoya, Aich, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sato Y, Shimizu S, Ueda K, Suzuki T, Suzuki S, Miura R, Ando M, Tsuda K, Iwata O, Muramatsu Y, Kidokoro H, Hirakawa A, Hayakawa M; SHEILD team. Safety and tolerability of a Muse cell-based product in neonatal hypoxic-ischemic encephalopathy with therapeutic hypothermia (SHIELD trial). Stem Cells Transl Med. 2024 Nov 12;13(11):1053-1066. doi: 10.1093/stcltm/szae071. PMID 39401019
- [Derived] Matsuyama N, Shimizu S, Ueda K, Suzuki T, Suzuki S, Miura R, Katayama A, Ando M, Mizuno M, Hirakawa A, Hayakawa M, Sato Y. Safety and tolerability of a multilineage-differentiating stress-enduring cell-based product in neonatal hypoxic-ischaemic encephalopathy with therapeutic hypothermia (SHIELD trial): a clinical trial protocol open-label, non-randomised, dose-escalation trial. BMJ Open. 2022 Apr 26;12(4):e057073. doi: 10.1136/bmjopen-2021-057073. PMID 35473726